CLINICAL TRIAL: NCT02727881
Title: OHR-1601: A Phase III Study of the Efficacy and Safety of Squalamine Lactate Ophthalmic Solution, 0.2% Twice Daily in Subjects With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Efficacy and Safety Study of Squalamine Ophthalmic Solution in Subjects With Neovascular AMD
Acronym: MAKO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ohr Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHR-1601
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD, CNV, choroidal neovascularization, retinal eye disease
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Exercise; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Squalamine solution, 0.2% BID (Experimental): Squalamine lactate ophthalmic solution, 0.2% bis in die (BID) + ranibizumab every 4 weeks
  Interventions: Drug: Squalamine lactate ophthalmic solution, 0.2%; Drug: ranibizumab
- Placebo solution BID (Placebo Comparator): Placebo ophthalmic solution BID + ranibizumab every 4 weeks
  Interventions: Drug: Placebo Ophthalmic solution; Drug: ranibizumab

INTERVENTIONS:
Drug: Squalamine lactate ophthalmic solution, 0.2% — Squalamine lactate ophthalmic solution, 0.2%
  Other Names: active
  Arms: Squalamine solution, 0.2% BID
Drug: Placebo Ophthalmic solution — Placebo Ophthalmic solution
  Other Names: placebo
  Arms: Placebo solution BID
Drug: ranibizumab — ranibizumab
  Other Names: Lucentis

SUMMARY:
A Phase 3 Study of the Efficacy and Safety of Squalamine Lactate Ophthalmic Solution 0.2% Twice Daily in Subjects with Neovascular Age-Related Macular Degeneration. Patients will receive injections of ranibizumab. In addition, patients will receive either Squalamine lactate 0.2% eye drops or Placebo eye drops. The study duration is approximately 9 months to primary endpoint

DETAILED DESCRIPTION:
Phase 3 Study of the Efficacy and Safety of Squalamine Lactate Ophthalmic Solution 0.2% Twice Daily in Subjects with Neovascular Age-Related Macular Degeneration Methodology: Phase III, multicenter, randomized, double-masked, placebo-controlled study conducted over 9 months

(Screening/Baseline to Week 36): Patients will be randomly assigned to one of 2 treatment groups in a 1:1 ratio:

* Squalamine lactate ophthalmic solution, 0.2% BID + ranibizumab every 4 weeks
* Placebo ophthalmic solution BID + monthly ranibizumab every 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* A diagnosis of choroid neovascularization (CNV) secondary to AMD with CNV comprising at least 50% of the total lesion area on fluorescein angiography (FA)
* Central subfield thickness (spectral domain (SD)-OCT central 1 mm) of ≥ 300 μm
* Best-corrected visual acuity (BCVA) 20/40 to 20/320 (73- to 24-letter score on the Early Treatment of Diabetic Retinopathy Study [ETDRS] chart)

Exclusion Criteria:

* Neovascularization secondary to any other condition than AMD in the study eye; Blood occupying greater than 50% of the AMD lesion, or blood > 1.0 sq. mm underlying the fovea
* Pigment epithelial detachment (PED) without associated subretinal fluid and/or cystic retinal changes
* Clinical evidence of diabetic retinopathy or diabetic macular edema in the study eye
* Confounding ocular conditions in the study eye which will affect interpretation of OCT, VA or assessment of macular appearance (e.g., cataract, epiretinal membrane, retinal vascular occlusive disease)
* Fibrosis or atrophy, retinal epithelial tear in the center of the fovea in the study eye or any condition preventing VA improvement
* Uncontrolled glaucoma in the study eye, or currently receiving topical glaucoma medication in the study eye

Ages: 50 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Functional change in visual acuity | 9 months
  Effect of combination therapy of ranibizumab monthly intravitreal injections with Squalamine Lactate Ophthalmic Solution, 0.2% on change in visual function as assessed by ETDRS BCVA in subjects with Age-Related Macular Degeneration

SECONDARY OUTCOMES:
Functional changes in visual acuity | 9 months
  Effect of combination therapy of ranibizumab monthly intravitreal injections with Squalamine Lactate Ophthalmic Solution, 0.2% on change in visual function as assessed by ETDRS BCVA in subjects with Age-Related Macular Degeneration

OTHER OUTCOMES:
Treatment emergent Adverse Event (AE) monitoring | 9 months
  Adverse and Serious Adverse Events in subjects receiving combination therapy of ranibizumab intravitreal injections with Squalamine Lactate Ophthalmic Solution, 0.2% assessed by adverse event reporting and Ophthalmic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Avner Ingerman, MD, Study Director — Ohr Pharmaceutical
Locations (109):
- United States (109):
  - Investigational Site, Mobile, Alabama
  - Investigational Site, Phoenix, Arizona
  - Investigational Site, Tucson, Arizona
  - Investigational Site, Arcadia, California
  - Investigational Site, Beverly Hills, California
  - Investigational Site, Campbell, California
  - Investigational Site, Fullerton, California
  - Investigational Site, Glendale, California
  - Investigational Site, Glendora, California
  - Investigational Site, La Jolla, California
  - Investigational Site, Laguna Hills, California
  - Investigational Site, Loma Linda, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, Oceanside, California
  - Investigational Site, Orange, California
  - Investigational Site, Palm Desert, California
  - Investigational Site, Palo Alto, California
  - Investigational Site, Pasadena, California
  - Investigational Site, Poway, California
  - Investigational Site, Redlands, California
  - Investigational Site, Sacramento, California
  - Investigational Site, Bridgeport, Connecticut
  - Investigational Site, Hamden, Connecticut
  - Investigational Site, New London, Connecticut
  - Investigational Site, Altamonte Springs, Florida
  - Investigational Site, Boynton Beach, Florida
  - Investigational Site, Fort Myers, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Naples, Florida
  - Investigational Site, Sarasota, Florida
  - Investigational Site, Stuart, Florida
  - Investigational Site, Augusta, Georgia
  - Investigational Site, ‘Aiea, Hawaii
  - Investigational Site, Berwyn, Illinois
  - Investigational Site, Bloomington, Illinois
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Sycamore, Illinois
  - Investigational Site, New Albany, Indiana
  - Investigational Site, Leawood, Kansas
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Paducah, Kentucky
  - Investigational Site, Portland, Maine
  - Investigational Site, Baltimore, Maryland
  - Investigational Site, Glen Burnie, Maryland
  - Investigational Site, Hagerstown, Maryland
  - Investigational Site, Pikesville, Maryland
  - Investigational Site, Rockville, Maryland
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Grand Rapids, Michigan
  - Investigational Site, Jackson, Michigan
  - Investigational Site, Royal Oak, Michigan
  - Investigational Site, Southfield, Michigan
  - Investigational Site, Traverse City, Michigan
  - Investigational Site, Biloxi, Mississippi
  - Investigational Site, Chesterfield, Missouri
  - Investigational Site, Florissant, Missouri
  - Investigational Site, Henderson, Nevada
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, Portsmouth, New Hampshire
  - Investigational Site, Bloomfield, New Jersey
  - Investigational Site, Lawrenceville, New Jersey
  - Investigational Site, New Brunswick, New Jersey
  - Investigational Site, Northfield, New Jersey
  - Investigational Site, Ramsey, New Jersey
  - Investigational Site, Teaneck, New Jersey
  - Investigational Site, Toms River, New Jersey
  - Investigational Site, Brooklyn, New York
  - Investigational Site, Great Neck, New York
  - Investigational Site, Hauppauge, New York
  - Investigational Site, Lynbrook, New York
  - Investigational Site, New York, New York
  - Investigational Site, Rochester, New York
  - Investigational Site, Rockville Centre, New York
  - Investigational Site, Syracuse, New York
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Concord, North Carolina
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Toledo, Ohio
  - Investigational Site, Youngstown, Ohio
  - Investigational Site, Ashland, Oregon
  - Investigational Site, Camp Hill, Pennsylvania
  - Investigational Site, Kingston, Pennsylvania
  - Investigational Site, Lancaster, Pennsylvania
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, Columbia, South Carolina
  - Investigational Site, Greenville, South Carolina
  - Investigational Site, Mt. Pleasant, South Carolina
  - Investigational Site, Rapid City, South Dakota
  - Investigational Site, Kingsport, Tennessee
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Fort Worth, Texas
  - Investigational Site, Grapevine, Texas
  - Investigational Site, Harlingen, Texas
  - Investigational Site, Houston, Texas
  - Investigational Site, Katy, Texas
  - Investigational Site, Kingwood, Texas
  - Investigational Site, McAllen, Texas
  - Investigational Site, Plano, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, The Woodlands, Texas
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Burlington, Vermont
  - Investigational Site, Fairfax, Virginia
  - Investigational Site, Warrenton, Virginia
  - Investigational Site, Bellevue, Washington
  - Investigational Site, Spokane, Washington
  - Investigational Site, Morgantown, West Virginia
  - Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No